CLINICAL TRIAL: NCT06839183
Title: Develop and Evaluate the Effectiveness of Integrated Interactive Self-care APP on Self-efficacy, Self-compassion and Resilience Among Patients Undergoing Hematopoietic Stem Cell Transplantation(the Second and Third-year Mixed-method Study)
Brief Title: Develop and Evaluate of Integrated Interactive Self-care APP Among Hematopoietic Stem Cell Transplantation Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KMUHIRB-F(I)20210187; MOST-111-2410-H-037-012 (Other Grant/Funding Number: Ministry of Science and Technology in Taiwan)
Record Dates: First submitted 2024-12-18; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-11

CONDITIONS: Mobile Health; Application; Hematopoietic Stem Cell Transplantations; Self-compassion; Resilience; Self Efficacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Application group (Experimental): use the integrated interactive self-care APP
  Interventions: Device: integrated interactive self-care APP
- usual care group (No Intervention): usual care

INTERVENTIONS:
Device: integrated interactive self-care APP — integrated interactive self-care APP
  Arms: Application group

SUMMARY:
Background: More than 50,000 hematopoietic stem cell transplants are performed around the world every year. However, HSCT treatment time is long and the treatment methods are complex, and it has a significant impact on the patient's body and mind. Foreign studies have shown that using mobile technology for cancer symptom monitoring and self-care can effectively improve cancer patients' doctor-patient communication, symptom management, and self-care abilities. There are only 7 articles on foreign HSCT-related APPs or online smart projects.

Purpose: To evaluate the use of an integrated interactive self-care APP in hematopoietic stem cell transplant patients Methods: This study is a two-stage explanatory qualitative mixed study. The quantitative study in the second year adopts a non-randomized experimental research design. Pre-test and formal testing are repeated in two groups. The experimental group (APP) will be admitted first according to the patient's wishes. The number of participants will then be included in the control group. Each group is expected to receive 40 subjects. The experimental group will receive general routine care plus the use of an integrated interactive self-care APP. The control group will receive general routine care and will be filled out at 8-time points before and after transplantation. Self-efficacy, self-compassion, and resilience questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Conscious, over 20 years old, and able to communicate in Mandarin or Taiwanese dialect.
2. Diagnosed via pathology report with one of the following cancers: acute myeloid leukemia, acute lymphoblastic leukemia, non-Hodgkin lymphoma, or multiple myeloma.
3. Requires HSCT (Hematopoietic Stem Cell Transplantation) treatment.
4. Possesses a smartphone.

Exclusion Criteria:

* All mental disorders as classified in the DSM-IV.

Min Age: 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
self-efficacy | Transplant Day 0 (T1), Day 7 (T2), Day 14 (T3), Day 30 (T4), Day 60 (T5), Day 90 (T6), Day 120 (T7).
  Self-efficacy will be measured using the Strategies Used By People To Promote Health, SUPPH, a validated 29-item scale scored from 29 to 145, where higher scores indicate greater self-efficacy."
self-compassion | Transplant Day 0 (T1), Day 7 (T2), Day 14 (T3), Day 30 (T4), Day 60 (T5), Day 90 (T6), Day 120 (T7).
  Self-compassion will be measured using the Self-Compassion Scale (SCS), a validated 26-item questionnaire scored from 1 to 5, where higher scores indicate greater self-compassion.
resilience | Transplant Day 0 (T1), Day 7 (T2), Day 14 (T3), Day 30 (T4), Day 60 (T5), Day 90 (T6), Day 120 (T7).
  Resilience will be measured using the Resilience Scale 14 item (RS-14), a 14-item scale scored from 7 to 98, where higher scores indicate greater resilience.
Usability assessments | Immediately after app intervention.
  Usability will be measured using the System Usability Scale (SUS), a validated 10-item scale scored from 0 to 100, where higher scores indicate better usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan